CLINICAL TRIAL: NCT07404540
Title: Effect of β-alanine Supplementation and Training on Ergogenic Parameters and Plasma Metabolites in Untrained Young Adults: a Randomized, Placebo-controlled, Double-blind Trial
Brief Title: Effect of β-alanine Supplementation and Training on Ergogenic Measures and Plasma Metabolites in Untrained Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, David Csala, Principal Investigator, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 316-2406-1/KK15/2011
Record Dates: First submitted 2026-01-29; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Dietary Supplementation; Healthy Vollunteer
Keywords: β-alanine; Exercise training; Dietary supplementation; Physical performance; Untrained adults

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to receive either β-alanine supplementation or a matchin
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- β-Alanine Supplementation (Experimental): Participants received β-alanine supplementation at a dose of 50 mg/kg/day, divided into multiple daily doses, in combination with a supervised six-week exercise training program.
  Interventions: Dietary Supplement: β-Alanine
- Placebo (Placebo Comparator): Participants received a visually identical placebo following the same dosing schedule as the supplementation group, in combination with a supervised six-week exercise training program.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: β-Alanine — β-alanine was administered orally at a dose of 50 mg/kg/day, divided into multiple daily doses and consumed with meals, throughout the six-week training intervention.
  Arms: β-Alanine Supplementation
Dietary Supplement: Placebo — Participants received visually identical placebo capsules following the same dosing schedule as the β-alanine group during the six-week training intervention.
  Arms: Placebo

SUMMARY:
This study enrolled untrained young adults to evaluate the effects of β-alanine supplementation combined with a structured exercise training program. Participants were randomly assigned to receive either β-alanine or a placebo while completing a six-week training regimen. Before and after the intervention, physical performance tests and blood samples were collected to assess changes in performance measures and biochemical markers in the blood. The purpose of the study was to determine how β-alanine supplementation influences exercise performance and related physiological outcomes in individuals who had not previously engaged in regular training.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled study was conducted to evaluate the effects of β-alanine supplementation combined with a structured exercise training program in untrained young adults. Participants were randomly assigned to receive either β-alanine supplementation or a matching placebo while completing a six-week supervised training intervention. Both participants and investigators responsible for training supervision and outcome assessments were blinded to group allocation.

The primary outcome measures focused on changes in physical performance capacity. Maximal muscle strength was assessed using standardized dynamometric measurements, and aerobic capacity was evaluated using a validated shuttle run test performed before and after the intervention.

Secondary outcome measures included changes in anthropometric parameters, pulmonary function, and exercise-related metabolic responses. Blood lactate concentrations were measured during standardized exercise testing to characterize metabolic responses to training and supplementation. In addition, fasting venous blood samples were collected before and after the intervention to determine plasma concentrations of β-alanine, histidine, and carnosine as biochemical outcome measures related to supplementation and training adaptation.

All outcome measures were collected at baseline and following completion of the six-week intervention period. Adverse events were monitored throughout the study duration through participant self-report and investigator observation. All study procedures were performed in accordance with ethical approval and institutional guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults aged 18-30 years.
* Untrained individuals without participation in structured resistance or endurance training during the previous 6 months.
* Not physically inactive, but not engaged in regular structured exercise training.
* Ability to participate in a six-week supervised multicomponent exercise training program.
* Willingness to comply with study procedures, training sessions, and supplementation protocol.
* Provision of written informed consent.

Exclusion Criteria:

* Known cardiovascular, metabolic, neuromuscular, or musculoskeletal disease.
* Acute injury at the time of enrollment.
* Regular use of medications or dietary supplements affecting muscle metabolism or exercise performance.
* Participation in structured resistance or endurance training during the previous 6 months.
* Failure to comply with the study protocol or training requirements.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in maximal muscle strength | Baseline and 6 weeks
  Maximal muscle strength was assessed by dynamometric measurements of maximal voluntary isometric contraction.
Change in aerobic capacity | Baseline and 6 weeks
  Aerobic capacity was estimated by VO₂max derived from the 20-m multistage fitness test (shuttle run).

SECONDARY OUTCOMES:
Body mass index (BMI) | Baseline and 6 weeks
  Body mass index calculated from measured height and body mass..
Body fat percentage | Baseline and 6 weeks
  Body fat percentage estimated from standardized skinfold thickness measurements.
Forced vital capacity (FVC) | Baseline and 6 weeks
  Forced vital capacity measured by spirometry using a portable spirometer to assess respiratory function.
Acute blood lactate response to dynamometric exercise | Baseline and 6 weeks
  Acute blood lactate responses were measured during standardized dynamometric exercise testing.
Plasma β-alanine concentration | Baseline and 6 weeks
  Plasma β-alanine concentration measured from fasting venous blood samples.
Plasma histidine concentration | Baseline and 6 weeks
  Plasma histidine concentration measured from fasting venous blood samples.
Plasma carnosine concentration | Baseline and 6 weeks
  Plasma carnosine concentration measured from fasting venous blood samples.

OTHER OUTCOMES:
Adverse events | Up to 6 weeks
  Adverse events monitored through participant self-report and investigator observation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly due to data protection and privacy considerations. De-identified data may be made available upon reasonable request to the corresponding author, subject to institutional approval.